CLINICAL TRIAL: NCT03674203
Title: Efficacy of Platelet-rich Plasma in Treatment of Melasma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, CLOTILDE FUENTES OROZCO, PhD, Instituto Mexicano del Seguro Social
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-2015-1301-88.
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Melasma
Keywords: Platelet-rich plasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: A prospective cohort study with therapeutic intervention for one year. We included patients older than 18 years with a diagnosis of melanoma and a history of pregnancy with a time greater than 6 months, who were not in the period of lactation, with no history of skin cancer, with a history of liver, thyroid or injury, of acne and traumatic injuries on the face, in addition, with no work history of PRP. The patients received three sessions of PRP application, at intervals of 15 days between each of them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Application of platelet-rich plasma (Experimental): The patients received three sessions of PRP application, at intervals of 15 days between each of them. It was applied by means of a 32G needle to introduce the PRP by means of superficial micro-injections via the mesotherapy technique (approximately 1.5-2.0 mm deep) and it was deposited in the papillary dermis of the rosotro.
  Interventions: Biological: Platelet-Rich Plasma

INTERVENTIONS:
Biological: Platelet-Rich Plasma — 1 ml of PRP was distributed in the papillary dermis of the face, repeating the dose at 15 and 30 days.

SUMMARY:
The application of Platelet Rich Plasma (PRP) on three occasions with an interval of 15 days between each one, is related to a decrease in the intensity of the spots and improvement in the quality of the skin of patients with melasma.

DETAILED DESCRIPTION:
832/5000 Objective: To evaluate the effect of PRP for Melasma treatment. Material and methods: Prospective cohort with therapeutic intervention. Patients, female, with melasma were included. Changes in the melanin concentration of the face (MASI), degree of satisfaction (MELASQOL) and histological changes were clinically evaluated.

The Sp-MELASQOL questionnaire, Fitzpatrick and MASI scales were applied, and photographs were taken with ambient light and with Wood's light with the Janus-II General Model. The patients were evaluated and classified, before and after the treatment by means of dermatoscopy, which was performed using a dermatoscope with polarized light (DermLite DL3N®), which allows an increase from 6 to 400X.

The dermatoscopy reported the findings of: Quantity, Density and Depth of melasma.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of melasma
* History of pregnancy with a time greater than 6 months
* Informed consent

Exclusion Criteria:

* In lactation period
* History of skin cancer
* History of liver, thyroid diseases
* With active acne lesions and traumatic lesions on the face
* PRP pre-treatmentPre-treatment for melasma with less than 6 months
* Hb values <10 g / dL or platelet count <105x109 / L

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change of the severity of melasma. | one year
  First divide the face into four regions: front (F), right malar (MR), left malar (ML), and chin (CH), which corresponds to 30%, 30%, 30% and 10% , respectively, of the total area(A) of the face. Subsequently, the area involved in each region is evaluated, assigning values from 1 to 6, depending on whether it affects: less than 10%; 10 to 29%; 30 to 49%; 50 to 69%; 70 to 89%; or 90 to 100%. A score is also assigned according to the darkening of the pigmentation (D): absent (0); mild (1); moderate (2); marked (3) or maximum (4). Finally, following this same scale, a value is assigned according to the homogeneity of the pigmentation (H).
  The following equation is used to calculate this index:
  The Melasma Area and Severity Index= 0.3 (DF + HF) AF+ 0.3 (DMR + HMR) AMR + 0.3 (DML + HML) AML + 0.1 (DCH + HCH) ACH
  The range is 0-48, although it is strictly an aesthetic problem, the higher the score, the greater the affectation. This scale was applied before and after the treatment.
Comparison of histological analysis | one year
  For this analysis, the obtained samples were fixed by 10% formalin and cuts of 6 μm were made. Hematoxylin-eosin staining was used for the visualization of melanophages in the dermis, cutaneous atrophy, solar elastosis and inflammatory infiltrate. Fontana-Masson stain to evaluate the pigmentation, focality of the pigmentation, distribution and absence of pigment in the papillary dermis.
  Biopsy was taken at the beginning of the study and at the end.
Type of melasma by dermatoscopy | one year
  It was performed using a dermatoscope (DermLite DL3N brand) with polarized light. Pictures were taken, (with Canon Powershot G12 camera) of the most characteristic part of the lesion, either in front, cheekbones or jaw. The photograph was taken before and after starting the treatment of the same anatomical site on both occasions. The melasma was classified according to the depth in: epidermal (regular and brown pigment is appreciated), dermal (regularity is lost and a color between blue and gray is seen) and mixed (combinations of these two). Two researchers were in charge of performing the dermatoscopy and the qualitative measurement of it.
Amount of melasma by dermatoscopy | one year
  Photographs were compared by dermatoscopy of the most characteristic part of the lesion before and after treatment. Categorizing these photographs in: 0 (without appreciable lesions), 1 (discolorations and slight presence of pigment), 2 (scattered pigment points) and 3 (pigment points together).
Density of melasma by dermatoscopy | one year
  Photographs were compared by dermatoscopy of the most characteristic part of the lesion before and after treatment. Categorizing these photographs in: 1 (brown pigment), 2 (gray-blue) or 3 (dark brown / black).
Presence or not of telangiectasias. | one year
  Photographs were compared by dermatoscopy of the most characteristic part of the lesion before and after treatment. In search of telangiectasias. Two researchers were in charge of performing the dermatoscopy and the qualitative measurement of it.

SECONDARY OUTCOMES:
change in the quality of life: Sp-MELASQOL | one year
  Melasma Quality of Life scale (MELASQOL) is a useful and objective tool to assess the quality of life of patients. In this protocol, the Sp-MELASQOL will be used, since it is the version in Spanish validated by Domínguez and cols, for the Latin American population. Which consists of 10 questions, with a score for each question from 1 to 7 points, where 1 = never and 7 = always.
  The results range from 7-70 points, the higher the score indicated, the lower the quality of life presented by the patients.
  We compare the results obtained before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde Fuentes, pHD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Western Medical Center, Mexican Institute of Social Security, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided